CLINICAL TRIAL: NCT04256408
Title: Bronchoscopic Conversion of Collateral Ventilation in CV-positive Emphysema Patients Before Endobronchial Valve Treatment - Mind The Gap Crossing Borders Study
Brief Title: Mind The Gap - Crossing Borders Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Pulmonx Corporation (Industry)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, Prof. dr. D.J. Slebos MD, PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mind The Gap
Record Dates: First submitted 2020-01-20; First posted 2020-02-05 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Emphysema; COPD; Hyperinflation Lung
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Treatment group
  Interventions: Device: Bronchoscopic transparenchymal interlobar fissure closure using Aeriseal

INTERVENTIONS:
Device: Bronchoscopic transparenchymal interlobar fissure closure using Aeriseal — Transbronchial or transparenchymal injection of AeriSeal into the interlobar collateral ventilation channels region to convert CV-positive lobes into CV-negative lobes.
  Other Names: Aeriseal

SUMMARY:
Rationale: A big step forward and great opportunity to improve overall efficacy of bronchoscopic lung volume reductioen is to combine treatment modalities aiming to close the dependent collateral channels and then proceed with EBV therapy to induce lobar collapse, and thus maximal treatment effect.

Objective:

Primary objective:

1. To investigate the feasibility of injecting AeriSeal into the interlobar collateral ventilation channels region to make the target lobe suitable for endobronchial valve treatment.

   Secondary objectives:
2. To investigate the safety of injecting AeriSeal into the interlobar collateral ventilation channels region to make the target lobe suitable for endobronchial valve treatment.
3. To investigate the effectiveness of injecting AeriSeal into the interlobar collateral ventilation channels region to make the target lobe suitable for endobronchial valve treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of emphysema with a treatable target for endobronchial valves (Zephyr).
2. Subjects of both genders of at least 35 years of age at the time of the baseline visit.
3. Understand and voluntarily sign a patient informed consent form.
4. 15 % predicted ≤ FEV1 ≤ 50% predicted.
5. RV ≥ 175% predicted, and TLC ≥ 100% predicted and RV/TLC ≥ 55%.
6. 6MWD ≥ 140 meters.
7. Dyspnea score of ≥2 on the mMRC scale of 0-4.
8. Non-smoker > 6 months prior to signing the informed consent.
9. Chartis CV positive between target and ipsilateral lobe

Exclusion Criteria:

1. Evidence of active pulmonary infection.
2. Evidence of clinically significant bronchiectasis.
3. History of more than 3 exacerbations with hospitalizations over the past 12 months.
4. Myocardial infarction or other relevant cardiovascular events in the past 6 months.
5. Prior lung surgery, Lung volume reduction surgery, lung transplantation, lobectomy, or pneumonectomy.
6. Prior endoscopic lung volume reduction.
7. Unstable pulmonary nodule requiring follow-up
8. Pregnant of nursing women.
9. Hypercapnia defined by PaCO2 > 8.0kPa, or Hypoxemia defined by PaO2 < 6.0kPa, both measured on room air.
10. Any disease with high probability of mortality within 24 months.
11. Patient is on an antiplatelet agent (such as Plavix) or anticoagulant therapy (such as LMWH or coumarins), which cannot be stopped periprocedural.
12. Patient was involved in other pulmonary drug studies within 30 days prior to this study.

    -

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
feasibility - Target Lobar Volume Change on Chest -CT scan | 3 months
  To investigate the feasibility of injecting AeriSeal into the interlobar collateral ventilation channels region to make the target lobe suitable for endobronchial valve treatment

SECONDARY OUTCOMES:
safety - Number and specification of reported (S)AEs per individual patient and as aggregate | 3 months
  To investigate the safety of injecting AeriSeal into the interlobar collateral ventilation channels region to make the target lobe suitable for endobronchial valve treatment. Thsi by collection of all adverse events, and specifically: death, pnuemothorax, pneumonia, COPD exacerbation, and post treatment inflammatory response.
changes in Quality of Life as measured by the SGRQ | 3 months
  By measuring the absolute change in The St George's Respiratory Questionnaire total score (0-100 points with higher scores indicating poor QOL)
effectiveness - Measurement of change in Forced Expiratory Volume in one second (FEV1). | 3 months
  By measuring changes in relative% in FEV1(L)
effectiveness - Measurement of change in Residual Volume (RV) | 3 months
  By measuring the change in absolute mL in RV
effectiveness - Measurement of changes in 6-minute walk test (6MWT) | 3 months
  By measuring the absolute change in meters in the 6MWT
changes in Quality of Life as measured by the COPD Assessment Test (CAT) | 3 months
  By measuring the absolute change in CAT score (0-40, with higher score indicating poor QOL)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Klooster, PhD, Study Director — UMC-Groningen/NL
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No